CLINICAL TRIAL: NCT01925014
Title: A Multi-institutional Trial Comparing Clinical Outcomes Following Low- vs. Standard-dose Abdominal CT as the First-line Imaging Test in Adolescents and Young Adults With Suspected Acute Appendicitis
Brief Title: Low vs. Standard Dose CT for Appendicitis Trial
Acronym: LOCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyoung Ho Lee, MD (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Seoul National University Bundang Hospital (Other); Radiology Imaging Network of Korea for Clinical Research (Other); The LOCAT Group (Unknown)
Responsible Party: Sponsor-Investigator, Kyoung Ho Lee, MD, Professor, Seoul National University Bundang Hospital
Organization: Seoul National University Bundang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LOCAT
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Appendicitis
Keywords: Appendectomy; Appendicitis; False Positive Reactions; Humans; Radiation Dosage; Tomography, X-Ray Computed; Young Adult
MeSH Terms: conditions — Appendicitis | interventions — Radiation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose CT (Experimental): Diagnostic CT with low-dose radiation
  Interventions: Diagnostic Test: Diagnostic CT with low-dose radiation
- Standard-dose CT (Active Comparator): Diagnostic CT with standard-dose radiation
  Interventions: Diagnostic Test: Diagnostic CT with standard-dose radiation

INTERVENTIONS:
Diagnostic Test: Diagnostic CT with low-dose radiation — Effective dose is aimed at approximately 2 millisievert (mSv) in an average patient.
  Other Names: Low-dose CT
  Arms: Low-dose CT
Diagnostic Test: Diagnostic CT with standard-dose radiation — Effective dose is aimed at approximately 8 millisievert (or less) in an average patient.
  Other Names: Standard-dose CT
  Arms: Standard-dose CT

SUMMARY:
To determine whether low-dose (LD) CT is noninferior to standard-dose (SD) computed tomography (CT) as the first-line imaging test in adolescents and young adults in regard to negative appendectomy rate (NAR).

DETAILED DESCRIPTION:
* Acute appendicitis is a very common disease. Many patients are adolescents or young adults.
* CT is the current standard imaging test for the diagnosis of appendicitis.
* In recent years, the awareness of carcinogenic risk associated with CT radiation has increased.
* According to a recent single-institutional randomized controlled trial, LD CT (employing a quarter of standard radiation dose) was found to be noninferior to SD CT with respect to NARs in adolescents and young adults with suspected appendicitis.
* However, LD CT is not yet widely accepted.
* To establish LD CT as the first-line imaging test, a multi-institutional study is needed to confirm the generalizability of the prior single-institutional study.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department visit with suspected symptoms and signs of acute appendicitis
* Intravenous contrast-enhanced computed tomography examination requested due to suspicion of appendicitis
* Willing to provide telephone or cell phone numbers for follow-up
* Signed informed consent provided prior to study entry

Exclusion Criteria:

* Prior cross-sectional imaging tests to evaluate the presenting symptoms and signs
* Prior history of surgical removal of the appendix

Ages: 15 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3074 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Ho Lee, MD, Study Chair — Seoul National University Bundang Hospital; Kyuseok Kim, MD, Study Director — Seoul National University Bundang Hospital
Locations (20):
- South Korea (20):
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Wonkwang University Sanbon Hospital, Sanbon, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Daejin Medical Center, Bundang Jesaeng General Hospital, Seongnam-si, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University School of Medicine & Hospital, Iksan
  - Gachon University Gil Medical Center, Incheon
  - Jeju National University Hospital, Jeju City
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, College of Medicine, Seoul St. Mary's Hospital, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Chung-Ang University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
The LOCAT Group has an active standpoint for sharing the LOCAT data, which is in line with the proposal from the International Committee of Medical Journal Editors. The LOCAT Group will share de-identified individual-participant data underlying the main LOCAT results no later than 6 months after the publication of the results. The data will be kept in a publicly available website and freely available to anyone upon request.

REFERENCES:
- [Background] Kim K, Kim YH, Kim SY, Kim S, Lee YJ, Kim KP, Lee HS, Ahn S, Kim T, Hwang SS, Song KJ, Kang SB, Kim DW, Park SH, Lee KH. Low-dose abdominal CT for evaluating suspected appendicitis. N Engl J Med. 2012 Apr 26;366(17):1596-605. doi: 10.1056/NEJMoa1110734. PMID 22533576
- [Background] Ahn S; LOCAT group. LOCAT (low-dose computed tomography for appendicitis trial) comparing clinical outcomes following low- vs standard-dose computed tomography as the first-line imaging test in adolescents and young adults with suspected acute appendicitis: study protocol for a randomized controlled trial. Trials. 2014 Jan 17;15:28. doi: 10.1186/1745-6215-15-28. PMID 24438500
- [Background] Ko Y, Choi JW, Kim DH, Lee KJ, Shin SS, Woo JY, Cho SW, Kim BS, Lee KH. Central image archiving and management system for multicenter clinical studies: lessons from low-dose CT for appendicitis trial. J Korean Soc Radiol. 2017 Mar 28;76(3):165-72. doi: 10.3348/jksr.2017.76.3.165.
- [Background] Yang HK, Ko Y, Lee MH, Woo H, Ahn S, Kim B, Pickhardt PJ, Kim MS, Park SB, Lee KH; Low-Dose CT for Appendicitis Trial (LOCAT) Group. Initial Performance of Radiologists and Radiology Residents in Interpreting Low-Dose (2-mSv) Appendiceal CT. AJR Am J Roentgenol. 2015 Dec;205(6):W594-611. doi: 10.2214/AJR.15.14513. PMID 26587949
- [Derived] Kim HY, Lee S, Kim DH, Ko Y, Park JH, Ko A, Jeong SM, Park SB, Lee KH; LOCAT Group. Conventional-Dose CT Versus 2-mSv CT for Right Colonic Diverticulitis as an Alternate Diagnosis of Appendicitis: Secondary Analysis of Large Pragmatic Randomized Trial Data. AJR Am J Roentgenol. 2021 Nov;217(5):1113-1121. doi: 10.2214/AJR.21.25584. Epub 2021 Apr 7. PMID 33825498
- [Derived] LOCAT Group. Low-dose CT for the diagnosis of appendicitis in adolescents and young adults (LOCAT): a pragmatic, multicentre, randomised controlled non-inferiority trial. Lancet Gastroenterol Hepatol. 2017 Nov;2(11):793-804. doi: 10.1016/S2468-1253(17)30247-9. Epub 2017 Sep 12. PMID 28919126
- See also: LOCAT-Training, a self-learning course to train the radiologists at all Sites to ensure the safety of the participants. — http://www.locat.org/locat_training

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 20 Korean teaching hospitals with predominantly limited experience in low-dose CT
Groups:
- Low-dose CT: 2 millisievert
- Standard-dose CT: 8 millisievert or lower
Period: Overall Study
Arm/Group | Low-dose CT | Standard-dose CT
Started | 1535 | 1539
Completed | 1526 | 1520
Not Completed | 9 | 19
Not completed — Inappropriate enrollment | 4 | 6
Not completed — Withdrawal by Subject | 5 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-dose CT | Standard-dose CT | Total
Number analyzed (Participants) | 1535 | 1539 | 3074
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Missing data due to withdrawal and inappropriate enrollment.
  years
    number analyzed (Participants) | 1526 | 1520 | 3046
    (all) | 28 [21 to 35] | 28 [21 to 35] | 28 [21 to 35]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Female | 838 | 834 | 1672
    Male | 688 | 686 | 1374
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    Ethnicity: number analyzed (Participants) | 1526 | 1520 | 3046
    Ethnicity: Korean | 1520 | 1504 | 3024
    Ethnicity: Non-Korean | 6 | 16 | 22
Body mass index (kg/m²) [Median (Inter-Quartile Range); unit: kg/m²] — Population: Missing data due to withdrawal and inappropriate enrollment.
  kg/m²
    number analyzed (Participants) | 1513 | 1505 | 3018
    (all) | 21.9 [19.8 to 24.5] | 22.1 [19.9 to 24.7] | 22.0 [19.8 to 24.6]
Body mass index (kg/m²) [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1513 | 1505 | 3018
    < 18.5 (underweight) | 151 | 147 | 298
    18.5-24.9 (normal) | 1044 | 1005 | 2049
    25.0-29.9 (overweight) | 268 | 292 | 560
    ≥ 30.0 (obese) | 50 | 61 | 111
Effective diameter (cm) [Median (Inter-Quartile Range); unit: cm] — The square root of the product of the anteroposterior diameter and lateral diameter of the abdomen, as measured on the transverse CT image at the umbilicus level. Population: Missing data due to withdrawal and inappropriate enrollment.
  cm
    number analyzed (Participants) | 1526 | 1520 | 3046
    (all) | 22.8 [20.7 to 25.2] | 22.8 [20.8 to 25.4] | 22.8 [20.8 to 25.3]
Effective diameter (cm) [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    < 20.0 | 227 | 242 | 469
    20.0-24.9 | 891 | 847 | 1738
    25.0-29.9 | 362 | 386 | 748
    ≥ 30.0 | 46 | 45 | 91
Chief complaint [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Abdominal pain | 1439 | 1439 | 2878
    Nausea/vomiting | 37 | 35 | 72
    Fever | 28 | 24 | 52
    Others | 22 | 22 | 44
Duration of symptoms [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    ≤ 12 hr | 606 | 621 | 1227
    13-24 hr | 402 | 430 | 832
    2-3 days | 381 | 354 | 735
    ≥ 4 days | 137 | 115 | 252
Location of abdominal pain [Count of Participants; unit: Participants] — Population: Patients may fall into more than one category. Missing data due to withdrawal and inappropriate enrollment.
  Participants
    Right lower quadrant: number analyzed (Participants) | 1526 | 1520 | 3046
    Right lower quadrant | 1344 | 1340 | 2684
    Suprapubic: number analyzed (Participants) | 1526 | 1520 | 3046
    Suprapubic | 228 | 204 | 432
    Right flank: number analyzed (Participants) | 1526 | 1520 | 3046
    Right flank | 209 | 190 | 399
    Periumbilical: number analyzed (Participants) | 1526 | 1520 | 3046
    Periumbilical | 172 | 173 | 345
    Epigastric: number analyzed (Participants) | 1526 | 1520 | 3046
    Epigastric | 156 | 118 | 274
    Other area(s): number analyzed (Participants) | 1526 | 1520 | 3046
    Other area(s) | 177 | 136 | 313
    No pain: number analyzed (Participants) | 1526 | 1520 | 3046
    No pain | 22 | 32 | 54
Migration of pain [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Yes | 466 | 452 | 918
    No | 1060 | 1068 | 2128
Abdominal tenderness [Count of Participants; unit: Participants] — Population: Patients may fall into more than one category. Missing data due to withdrawal and inappropriate enrollment.
  Participants
    Right lower quadrant: number analyzed (Participants) | 1526 | 1520 | 3046
    Right lower quadrant | 1305 | 1303 | 2608
    Epigastric: number analyzed (Participants) | 1526 | 1520 | 3046
    Epigastric | 147 | 151 | 298
    Left lower quadrant: number analyzed (Participants) | 1526 | 1520 | 3046
    Left lower quadrant | 124 | 97 | 221
    Suprapubic: number analyzed (Participants) | 1526 | 1520 | 3046
    Suprapubic | 112 | 115 | 227
    Periumbilical: number analyzed (Participants) | 1526 | 1520 | 3046
    Periumbilical | 104 | 129 | 233
    Other area(s): number analyzed (Participants) | 1526 | 1520 | 3046
    Other area(s) | 106 | 89 | 195
    No tenderness: number analyzed (Participants) | 1526 | 1520 | 3046
    No tenderness | 142 | 139 | 281
Rebound tenderness [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Yes | 634 | 570 | 1204
    No | 892 | 950 | 1842
Body temperature [Median (Inter-Quartile Range); unit: ℃] — Population: Missing data due to withdrawal and inappropriate enrollment.
  ℃
    number analyzed (Participants) | 1526 | 1520 | 3046
    (all) | 36.8 [36.5 to 37.2] | 36.8 [36.5 to 37.2] | 36.8 [36.5 to 37.2]
White blood cell (10³/mm³) [Median (Inter-Quartile Range); unit: 10³ cells/mm³] — Population: Missing data due to withdrawal and inappropriate enrollment.
  10³ cells/mm³
    number analyzed (Participants) | 1519 | 1513 | 3032
    (all) | 10.6 [7.8 to 13.6] | 10.6 [8.0 to 13.9] | 10.6 [7.9 to 13.8]
Segmented neutrophil (%) [Median (Inter-Quartile Range); unit: percentage of neutrophils] — Population: Missing data due to withdrawal and inappropriate enrollment.
  percentage of neutrophils
    number analyzed (Participants) | 1519 | 1512 | 3031
    (all) | 75 [64 to 82] | 75 [64 to 82] | 75 [64 to 82]
C-reactive protein (mg/dL) [Median (Inter-Quartile Range); unit: mg/dL] — Population: Missing data due to withdrawal and inappropriate enrollment.
  mg/dL
    number analyzed (Participants) | 1505 | 1504 | 3009
    (all) | 0.8 [0.2 to 3.5] | 0.7 [0.1 to 3.5] | 0.7 [0.1 to 3.5]
Alvarado score [Count of Participants; unit: Participants] — Alvarado score is a clinical scoring system used in the diagnosis of appendicitis. The score has 6 clinical items and 2 laboratory measurements with a total 10 points. A greater Alvarado score indicates a higher likelihood of appendicitis. Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1519 | 1512 | 3031
    Low risk (0-4) | 564 | 588 | 1152
    Indeterminate risk (5-8) | 864 | 836 | 1700
    High risk (9-10) | 91 | 88 | 179
Appendicitis inflammatory response score [Count of Participants; unit: Participants] — The appendicitis inflammatory response (AIR) score is a clinical scoring system used in the diagnosis of appendicitis. The score has 4 clinical items and 3 laboratory measurements with a total 12 points. A greater AIR score indicates a higher likelihood of appendicitis. Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1504 | 1503 | 3007
    Low risk (0-4) | 841 | 846 | 1687
    Indeterminate risk (5-8) | 643 | 624 | 1267
    High risk (9-12) | 20 | 33 | 53
Time of CT examination [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Working hours | 655 | 651 | 1306
    After hours | 871 | 869 | 1740
CT machine [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    16-channel | 301 | 300 | 601
    64-channel | 385 | 381 | 766
    128-channel | 568 | 567 | 1135
    256-channel | 272 | 272 | 544
Target effective dose (low-dose CT vs. standard-dose CT) [Count of Participants; unit: Participants] — While the effective dose for low-dose CT was aimed at 2 mSv for all CT machines, the target effective dose for standard-dose CT was individualized for each CT machine following the institutional normal dose. Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    2 mSv vs. 3 mSv | 25 | 23 | 48
    2 mSv vs. 5 mSv | 34 | 34 | 68
    2 mSv vs. 6 mSv | 398 | 396 | 794
    2 mSv vs. 7 mSv | 527 | 523 | 1050
    2 mSv vs. 8 mSv | 542 | 544 | 1086
Dose-length product (mGy·cm) [Median (Inter-Quartile Range); unit: mGy·cm] — Population: Missing data due to withdrawal and inappropriate enrollment.
  mGy·cm
    number analyzed (Participants) | 1525 | 1518 | 3043
    (all) | 132 [119 to 151] | 486 [390 to 561] | 274 [131 to 491]
Volume CT dose index (mGy) [Median (Inter-Quartile Range); unit: mGy] — Population: Missing data due to withdrawal and inappropriate enrollment.
  mGy
    number analyzed (Participants) | 1525 | 1518 | 3043
    (all) | 2.6 [2.2 to 2.7] | 9.4 [7.6 to 10.4] | 5.2 [2.6 to 9.4]
Size-specific dose estimate (mGy) [Median (Inter-Quartile Range); unit: mGy] — Population: Missing data due to withdrawal and inappropriate enrollment.
  mGy
    number analyzed (Participants) | 1525 | 1518 | 3043
    (all) | 4.1 [3.7 to 4.5] | 14.4 [12.9 to 16.2] | 9.1 [4.1 to 14.4]
Iterative reconstruction [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Used | 593 | 158 | 751
    Not used | 933 | 1362 | 2295
Radiologist who made initial CT report [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Attending radiologist | 886 | 863 | 1749
    On-call radiologist or trainees | 640 | 657 | 1297
Site characteristics: low-dose CT experience in the previous trial [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    Yes | 159 | 159 | 318
    No | 1367 | 1361 | 2728
Site characteristics: number of beds [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    < 650 | 363 | 360 | 723
    650-949 | 541 | 535 | 1076
    ≥ 950 | 622 | 625 | 1247
Site characteristics: annual number of appendectomies [Count of Participants; unit: Participants] — Population: Missing data due to withdrawal and inappropriate enrollment.
  Participants
    number analyzed (Participants) | 1526 | 1520 | 3046
    < 150 | 59 | 58 | 117
    150-299 | 329 | 323 | 652
    300-449 | 518 | 516 | 1034
    ≥ 450 | 620 | 623 | 1243

OUTCOME MEASURES:

1. Primary Outcome: Negative Appendectomy Rate
Description: Negative appendectomy rate was defined as the percentage of negative (unnecessary) appendectomies among all non-incidental appendectomies. As a secondary analysis, negative appendectomy rate in an alternative definition was calculated by excluding cases with appendiceal neoplasms without superimposed appendicitis, as appendectomy would be clinically necessary in such patients. Any surgery performed for the treatment of presumed appendicitis was counted as non-incidental appendectomy, even though the surgical procedures were more extensive than simple appendectomy (e.g., ileocectomy).
Time Frame: 1 week after surgery
Population: Patients who underwent appendectomy. Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 559 | 601
Participants
  Negative appendectomy (NA) rate | 22 | 16
  Not counting appendiceal neoplasm(s) as NA | 21 | 16
Statistical Analysis 1: Comparison: Low-dose CT vs Standard-dose CT; Detailed in Ahn S, LOCAT Group. Trials 2014:15:28; Test type: Non-Inferiority — Detailed in Ahn S, LOCAT Group. Trials 2014:15:28; Risk Difference (RD) = 0.013, 95% CI 2-sided [-0.008 to 0.033] — The non-inferiority was established

2. Secondary Outcome: Appendiceal Perforation Rate
Description: The percentage of perforated appendicitis among confirmed appendicitis cases.
Time Frame: 1 week after surgery
Population: Patients confirmed as having appendicitis. Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 524 | 564
Participants | 182 | 176
Statistical Analysis 1: Comparison: Low-dose CT vs Standard-dose CT; Detailed in Ahn S, LOCAT Group. Trials 2014:15:28; Test type: Non-Inferiority — Detailed in Ahn S, LOCAT Group. Trials 2014:15:28; Risk Difference (RD) = 0.035, 95% CI 2-sided [-0.021 to 0.091] — The non-inferiority was established

3. Secondary Outcome: Number of Appendectomies
Description: Appendectomy rate. The percentage of appendectomies among all randomized cases.
Time Frame: 3 months after CT
Population: Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Participants | 559 | 601

4. Secondary Outcome: Number of Negative Appendectomies
Description: The percentage of negative appendectomies among all randomized cases. In January, 2016, when more than 2000 patients were enrolled, the data and safety monitoring board noted a between-group imbalance in the number of appendectomies. Because of the concern that such an imbalance might potentially jeopardize the comparability for the prespecified endpoints, the study protocol was amended to adopt the following additional secondary endpoints, which were assessed among all randomly assigned patients: the number of appendectomies, number of negative appendectomies, prevalence of perforated appendicitis, and prevalence of non-perforated appendicitis.
Time Frame: 1 week after surgery
Population: Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Participants | 22 | 16

5. Secondary Outcome: Prevalence of Perforated Appendicitis
Description: The percentage (i.e., prevalence) of perforated appendicitis among all randomized cases. In January, 2016, when more than 2000 patients were enrolled, the data and safety monitoring board noted a between-group imbalance in the number of appendectomies. Because of the concern that such an imbalance might potentially jeopardize the comparability for the prespecified endpoints, the study protocol was amended to adopt the following additional secondary endpoints, which were assessed among all randomly assigned patients: the number of appendectomies, number of negative appendectomies, prevalence of perforated appendicitis, and prevalence of non-perforated appendicitis.
Time Frame: 1 week after surgery
Population: Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Participants | 182 | 176

6. Secondary Outcome: Prevalence of Non-perforated Appendicitis
Description: The percentage (i.e., prevalence) of non-perforated appendicitis among all randomized cases. In January, 2016, when more than 2000 patients were enrolled, the data and safety monitoring board noted a between-group imbalance in the number of appendectomies. Because of the concern that such an imbalance might potentially jeopardize the comparability for the prespecified endpoints, the study protocol was amended to adopt the following additional secondary endpoints, which were assessed among all randomly assigned patients: the number of appendectomies, number of negative appendectomies, prevalence of perforated appendicitis, and prevalence of non-perforated appendicitis.
Time Frame: 1 week after surgery
Population: Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Participants | 342 | 388

7. Secondary Outcome: Need for Additional Imaging Test(s)
Description: The proportion of patients requiring additional imaging test(s) in order to diagnose or rule out appendicitis.
Time Frame: 1 week after CT
Population: Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Participants | 39 | 41

8. Secondary Outcome: Delay in Patient Disposition
Description: * The interval from CT acquisition to appendectomy in patients undergoing appendectomy. Interval appendectomies following percutaneous abscess drainage and/or medical treatment were not included in this analysis.
  * The interval from CT acquisition to hospital discharge in patients not undergoing surgery.
Time Frame: 3 months after CT
Population: Intention-to-treat.
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1535 | 1539
Hours
  Interval between CT and appendectomy: number analyzed (Participants) | 535 | 589
  Interval between CT and appendectomy | 5.3 [3.1 to 9.7] | 5.4 [3.4 to 10.6]
  Interval between CT and discharge without surgery: number analyzed (Participants) | 936 | 875
  Interval between CT and discharge without surgery | 1.7 [0.9 to 3.9] | 1.6 [0.9 to 4.1]

9. Secondary Outcome: Length of Hospital Stay Associated With Appendectomy
Description: The interval from CT acquisition to hospital discharge after appendectomy.
Time Frame: 3 months after CT
Population: Patients who underwent appendectomy. Intention-to-treat. Interval appendectomies following percutaneous abscess drainage and/or medical treatment were not included in this analysis.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 538 | 590
Days | 3.0 [2.4 to 4.0] | 2.9 [2.2 to 3.9]

10. Secondary Outcome: Diagnostic Performance of CT Reports - AUC
Description: - Area under the receiver-operating-characteristic curve (AUC).
Time Frame: 3 months after CT
Population: Patients with incomplete reference standards were not included in these analyses. Intention-to-treat.
Measure: Number; unit: AUC
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1459 | 1429
AUC | 0.983 | 0.986

11. Secondary Outcome: Diagnostic Performance of CT Reports - Sensitivity and Specificity
Description: * Diagnostic sensitivity and specificity: the 5-grade likelihood scores for appendicitis were collapsed into binary responses with a decision threshold of a score ≥ 3 as positive for the diagnosis.
  * Sensitivity is a proportion of the positive test among the patient confirmed as having appendicitis.
  * Specificity is a proportion of the negative test among the patient confirmed as not having appendicitis.
Time Frame: 3 months after CT
Population: Patients with incomplete reference standards were not included in these analyses. Intention-to-treat.
Measure: Number; unit: percentage
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1459 | 1429
percentage
  Sensitivity (%): number analyzed (Participants) | 524 | 564
  Sensitivity (%) | 97.1 | 98.0
  Specificity (%): number analyzed (Participants) | 935 | 855
  Specificity (%) | 95.8 | 94.0

12. Secondary Outcome: Diagnostic Confidence in Diagnosing and Ruling Out Appendicitis: Likelihood Score for Appendicitis
Description: * Likelihood score for appendicitis in patients confirmed as having appendicitis.
  * Likelihood score for appendicitis in patients confirmed as not having appendicitis.
  Grade 1 denotes appendicitis definitely absent; grade 2, appendicitis probably absent; grade 3, indeterminate for the presence of appendicitis; grade 4, appendicitis probably present; and grade 5, appendicitis definitely present.
Time Frame: 3 months after CT
Population: Patients with incomplete reference standards were not included in these analyses. Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1459 | 1429
Participants
  Patients confirmed as having appendicitis: number analyzed (Participants) | 524 | 564
  Patients confirmed as having appendicitis: Grade 1 | 6 | 6
  Patients confirmed as having appendicitis: Grade 2 | 9 | 5
  Patients confirmed as having appendicitis: Grade 3 | 18 | 19
  Patients confirmed as having appendicitis: Grade 4 | 91 | 68
  Patients confirmed as having appendicitis: Grade 5 | 400 | 466
  Patients confirmed as not having appendicitis: number analyzed (Participants) | 935 | 865
  Patients confirmed as not having appendicitis: Grade 1 | 742 | 710
  Patients confirmed as not having appendicitis: Grade 2 | 154 | 103
  Patients confirmed as not having appendicitis: Grade 3 | 16 | 34
  Patients confirmed as not having appendicitis: Grade 4 | 14 | 10
  Patients confirmed as not having appendicitis: Grade 5 | 9 | 8

13. Secondary Outcome: Diagnostic Confidence in Diagnosing and Ruling Out Appendicitis: Indeterminate Interpretation (Grade 3)
Description: The frequency of indeterminate CT interpretation (grade 3). Grade 1 denotes appendicitis definitely absent; grade 2, appendicitis probably absent; grade 3, indeterminate for the presence of appendicitis; grade 4, appendicitis probably present; and grade 5, appendicitis definitely present.
Time Frame: 3 months after CT
Population: Patients with incomplete reference standards were not included in these analyses. Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 1459 | 1429
Participants | 34 | 53

14. Secondary Outcome: Diagnostic Confidence in Ruling Out Appendicitis: Normal Appendix Visualization
Description: The frequency of normal appendix visualization at CT. Grade 0 denotes appendix not identified; grade 1, unsure or partly visualized; and grade 2, clearly and entirely visualized.
Time Frame: 3 months after CT
Population: Patients confirmed as not having appendicitis. Intention-to-treat.
Measure: Count of Participants; unit: Participants
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 935 | 865
Participants
  Grade 0 | 36 | 14
  Grade 1 | 137 | 64
  Grade 2 | 762 | 787

15. Secondary Outcome: Diagnosis of Appendiceal Perforation at CT
Description: * Diagnostic sensitivity: the number of correct detections of the perforation divided by the number of cases of perforated appendicitis.
  * Diagnostic specificity: the number of correct ruling out the perforation divided by the number of cases of appendicitis without perforation.
Time Frame: 3 months after CT
Population: Patients confirmed to have appendicitis. Intention-to-treat.
Measure: Number; unit: Percentage
Arm/Group | Low-dose CT | Standard-dose CT
Number analyzed (Participants) | 524 | 564
Percentage
  Sensitivity (%): number analyzed (Participants) | 182 | 176
  Sensitivity (%) | 43 | 43
  Specificity (%): number analyzed (Participants) | 342 | 388
  Specificity (%) | 89 | 91

ADVERSE EVENTS:
Time Frame: 3 months
Description: Detailed in Ahn S, LOCAT Group. Trials 2014:15:28.
Arm/Group | Low-dose CT | Standard-dose CT
All-Cause Mortality (participants affected / at risk) | 0/1535 | 0/1539
Serious Adverse Events (participants affected / at risk) | 43/1535 | 40/1539
Other Adverse Events (participants affected / at risk) | 0/1535 | 0/1539
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-dose CT (N=1535) | Standard-dose CT (N=1539)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorders-other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 2 (2)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 4 (4) | 9 (9)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 4 (4) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Large intestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Surgical and medical procedures- other, specify (Surgical and medical procedures) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No